CLINICAL TRIAL: NCT06988150
Title: A Prospective Study to Assess the Prevalence of Small Intestinal Bacterial Overgrowth (SIBO) in Pancreatic Adenocarcinoma (PDAC) Patients With Weight Loss
Brief Title: Small Intestinal Bacterial Overgrowth (SIBO) in Pancreatic Adenocarcinoma (PDAC)
Acronym: SIBO in PDAC
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Hendifar, MD, Sponsor-Investigator, Cedars-Sinai Medical Center
Other Study IDs: STUDY00004075
Record Dates: First submitted 2025-04-23; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Adenocarcinoma; Weight Loss
Keywords: PDAC
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic adenocarcinoma with clinically significant weight loss.: Patients diagnosed with pancreatic adenocarcinoma with clinically significant weight loss.

SUMMARY:
The purpose of this study is to prospectively analyze the prevalence of SIBO in patients with Pancreatic adenocarcinoma (PDAC) and understand its association with weight loss and pancreatic resection status. Each patient will be tested for SIBO using Lactulose Hydrogen Breath Test. 100 patients with diagnosed pancreatic adenocarcinoma and clinically diagnosed weight loss will be enrolled in this study.

DETAILED DESCRIPTION:
Small intestinal bacterial overgrowth syndrome (SIBO) is a condition defined by excessive (greater than 105 CFU/mL) or abnormal bacteria in the upper gastrointestinal tract resulting in unintentional weight loss, diarrhea, nutritional deficiencies and osteoporosis. In healthy individuals, the growth of any remaining bacteria in the stomach is limited by biliary and pancreatic secretions. The location of Pancreatic ductal adenocarcinoma (PDAC) on the pancreas head hinders these exocrine secretions from reaching the small intestine, leading to exocrine pancreatic insufficiency in pancreatic cancer patients. Patients with Pancreatic adenocarcinoma suffer from similar symptoms including weight loss, diarrhea, and nutritional deficiencies. SIBO has been linked to Exocrine Pancreatic Insufficiency or anatomical abnormalities, both consistent in PDAC patients, especially those who have undergone surgery. Post-pancreatoduodenectomy physiological changes disrupt the way enzymes are secreted, which affects exocrine and endocrine functions of the pancreas. Currently, there is a limited understanding of the prevalence of SIBO in PDAC patients.

The primary objective of this study is to assess the prevalence of SIBO in consecutive PDAC patients with clinically significant weight loss.

The secondary objective of this study is to assess the prevalence of SIBO in patients who have undergone pancreatic resection versus those who have not undergone resection.

ELIGIBILITY:
Inclusion Criteria:

* Men, Women, and all genders
* Individuals 18 years old or older are included.
* Patients of the study investigators and team members
* Diagnosis of pancreatic ductal adenocarcinoma
* All subjects must consent to this study
* Clinically diagnosed weight loss

Exclusion Criteria:

* Minors
* Pregnant Women
* Any records flagged "break the glass" or "research opt out."
* Patients who have received treatment for SIBO in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pancreatic adenocarcinoma with clinically significant weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
SIBO in PDAC | At Screening Visit
  Assess the prevalence of SIBO in consecutive PDAC patients with clinically significant weight loss.

SECONDARY OUTCOMES:
SIBO & Resection | At Screening Visit
  Assess the prevalence of SIBO in patients who have undergone pancreatic resection versus those who have not undergone resection.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E. Hendifar, M.D., M.P.H., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No